CLINICAL TRIAL: NCT04766073
Title: Surgical Incision Closure Method to Prevent Niche Formation After Cesarean Section- Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8978006-HMO-CTIL
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Section Complications; Uterine Bleeding
MeSH Terms: conditions — Uterine Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Closure Technique (Experimental): This group will have the uterus closed after delivery of the fetus during cesarean section with a new technique.
  Interventions: Procedure: Niche prevention suture
- Regular closure technique (No Intervention): The usual method of closing the surgical incision is to suture the entire wall of the uterus with a stratafix suture without locking the suture.

INTERVENTIONS:
Procedure: Niche prevention suture — This group will have the uterus sutured in two layers using a new technique.
  Arms: New Closure Technique

SUMMARY:
In the last decade we have been exposed to the complication of a caesarean section called a "niche". A niche is an anaerobic defect in the location of the cesarean section, which represents the discontinuity of the endometrium and myometrium. A niche is usually diagnosed by ultrasound, and can also be diagnosed by hysterosalpingogram or hysteroscopy. In the presence of a niche women suffer more frequently from irregular bleeding, dysmenorrhea, chronic pelvic pain, and dyspareunia. We believe that a combination of tissue ischemia and thinning of the scar tissue that forms, causes a niche to form. Large randomized studies regarding the preferred surgical technique in cesarean section, including various methods of incision closure have found that there is no single method that is obviously superior. However, these studies did not examine niche formation as a complication of cesarean section.

In this study we will examine whether a unique incision closure method reduces post-cesarean niche formation.

ELIGIBILITY:
Inclusion Criteria:

* Women at first cesarean delivery
* Women who consent to the study

Exclusion Criteria:

* Women who are having a repeat caesarean section
* Refusal to participate in the study
* Urgent or emergent cesarean delivery

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 183 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Formation of a uterine niche | At least 12 weeks after delivery.
  Presence of a uterine niche on ultrasound

SECONDARY OUTCOMES:
Duration of surgery | At surgery
  Total duration of surgery
Blood loss over 1000 mL | At surgery
  As assessed by the operating surgeon
Postoperative infection | Up to 6 weeks after intervention
  The number of patients who are diagnosed with postoperative infection including endometritis or wound infection.
Need for repeat laparotomy | Up to 6 weeks after intervention
  The number of patients who undergo a repeat laparotomy after the initial cesarean delivery will be ascertained.
Formation of a n abscess/hematoma | Up to 6 weeks after intervention
  The number of patients who are diagnosed with a pelvic abscess or hematoma from the time of the cesarean delivery until 6 weeks after the cesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Hila Hochler, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No